CLINICAL TRIAL: NCT01115036
Title: Phase II Study of Panobinostat (LBH589) for Recurrent Glioblastoma (GBM) Undergoing Planned Surgical Resection
Brief Title: A Panobinostat Presurgery
Acronym: CLBH589C
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled on this study, so study was closed and IND withdrawn.
Sponsor: Duke University (Other)
Collaborators: Novartis (Industry)
Responsible Party: David A. Reardon, M.D., Preston Robert Tisch Brain Tumor Center at Duke University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020612
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2011-12

CONDITIONS: Recurrent Glioblastoma
Keywords: glioblastoma; recurrent; surgical resection
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- panobinostat (Experimental)
  Interventions: Drug: panobinostat

INTERVENTIONS:
Drug: panobinostat — Oral panobinostat will be administered at 20mg by mouth 3 times a week one week prior to surgical resection. Within 2-6 weeks of resection, patients will resume panobinostat at 20mg 3 times per week. A cycle will be 28 days.
  Other Names: LBH589

SUMMARY:
In the current study, the investigators will evaluate intratumoral pharmacodynamic and pharmacokinetic data associated with the administration of the HDACI, Panobinostat, among recurrent GBM patients. In addition, this study will evaluate the safety and tolerability of this agent, as well as evidence of anti-tumor activity in the patient population.

DETAILED DESCRIPTION:
This study will enroll a maximum of 24 subjects with recurrent GBM who are scheduled for planned debulking craniotomy.

After screening and enrollment on the study, subjects will receive 20mg panobinostat 3 times a week for one week prior to surgery. Within 2-6 weeks of resection, subjects will resume panobinostat at 20mg panobinostat 3 times per week.

The primary endpoint will be 6-month progression-free survival. Each cycle of therapy will be 28 days. All subjects will be assessed after every other cycle of therapy. Subjects will remain on study therapy for at least one year unless they develop progressive disease, unacceptable toxicity, non-compliance with study procedures or withdraw consent. Patients may continue treatment with oral panobinostat until they experience unacceptable toxicity that precludes further treatment, disease progression, and/or at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is ≥ 18 years
* Histologically-confirmed grade 4 malignant glioma patients;
* Candidate for surgical resection of tumor;
* No more than 3 prior episodes of progressive disease;
* An interval of at least 4 weeks between prior surgical resection or two weeks from stereotactic biopsy;
* An interval of at least 12 weeks from the end of prior radiotherapy unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there are progressive changes on MRI on at least two consecutive MRI scans at least four weeks apart, or there is biopsy-proven tumor progression;
* An interval of at least 4 weeks from prior chemotherapy (6 weeks for nitrosoureas) or investigational agent, unless the patient has recovered from all anticipated toxicities associated with that therapy;
* Karnofsky * 70%;
* Hemoglobin ≥ 9 g/dL, ANC > 1,500 cells/*l, platelets > 150,000 cells/*l ;
* Serum creatinine < 1.5 mg/dl or 24-hour creatinine clearance ≥ 50 ml/min, serum SGOT and bilirubin < 1.5 times upper limit of normal; total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN; serum potassium ≥ LLN; serum sodium ≥ LLN; serum albumin ≥ LLN or 3g/dl;
* Clinically euthyroid (Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism);
* Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal;
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed;

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment;
* Use of CYP-3A inducing anti-epileptics (phenytoin, fosphenytoin, carbamazepine, oxcarbazepine, phenobarbitol, primidone);
* Pregnancy or breast feeding;
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids;
* Active infection requiring intravenous antibiotics;
* Prior bevacizumab within 6 weeks of study enrollment;
* Therapeutic anti-coagulation with warfarin, aspirin, non-steroidal anti-inflammatory drugs or clopidogrel;
* Impaired cardiac function including any one of the following:

  * Complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (<50 beats per minute), QTcF > 450 msec on screening ECG, or right bundle branch block + left anterior hemiblock (bifascicular block);
  * Presence of atrial fibrillation (ventricular heart rate >100 bpm);
  * Previous history angina pectoris or acute MI within 6 months;
  * Congestive heart failure (New York Heart Association functional classification III-IV) or baseline MUGA/Echo shows LVEF < 45%;
* Uncontrolled hypertension;
* Concomitant use of drugs with a risk of causing Torsades de pointes (See Table 14-1);
* Patients with unresolved diarrhea ≥ grade 2;
* Patients with ≥ grade 2 peripheral neuropathy;
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
* Other concurrent severe and/or uncontrolled medical conditions;
* Concomitant use of any anti-cancer therapy or radiation therapy;
* Patients with a history of another primary malignancy within 5 years other than curatively treated carcinoma in situ of the cervix, or basal or squamous cell carcinoma of the skin;
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required;
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral panobinostat;
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Anti-tumor Activity as Measured by Percentage of Patients Who Remain Progression-free after Six Months | 18 months
  The primary objective will be to determine the anti-tumor activity of panobinostat among recurrent GBM patients as measured by the percentage of patients who remain progression-free after 6 months of therapy (PFS-6)

SECONDARY OUTCOMES:
Safety Evaluation of Panobinostat | 24 months
  A secondary objective is to further evaluate the safety of panobinostat in recurrent GBM patients
Evaluation of Intratumoral Pharmacokinetics and Pharmacodynamics of Panobinostat | 24 months
  A secondary objective is to evaluate the intratumoral pharmacokinetics and pharmacodynamics of panobinostat among recurrent GBM patients scheduled for surgical debulking
Evaluation of Systemic Pharmacokinetics | 24 months
  A secondary objective is to evaluate the systemic pharmacokinetics of panobinostat among recurrent GBM patients.

CONTACTS AND LOCATIONS:
Overall Officials: David A Reardon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States